CLINICAL TRIAL: NCT01926028
Title: Phase 1b/2a, Multi-center, Double-blind, Randomized, Placebo-controlled Study of a Single Dose of NDV-3A or NDV-3 Vaccine to Evaluate Safety, Tolerability, Immunogenicity and Efficacy in Preventing Recurrent Vulvovaginal Candidiasis
Brief Title: Safety, Tolerability, Immunogenicity and Efficacy of NDV-3A Vaccine in Preventing Recurrent Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NovaDigm Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NDV3A-003
Record Dates: First submitted 2013-08-09; First posted 2013-08-20 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Vulvovaginal Candidiasis
Keywords: recurrent vulvovaginal candidiasis; candida; NDV3; vaginal thrush; chronic yeast infection
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Torulopsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NDV-3A (Experimental): Experimental Vaccine: a purified, recombinant antigen (rAls3) formulated with aluminum hydroxide adjuvant
  Interventions: Biological: NDV-3A
- NDV-3 (Experimental): Experimental Vaccine: a purified, recombinant antigen (rAls3 with 6-His tag) formulated with aluminum hydroxide adjuvant
  Interventions: Biological: NDV-3
- Placebo (Placebo Comparator): Placebo: aluminum hydroxide adjuvant
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NDV-3A — 0.5mL injection IM
  Arms: NDV-3A
Biological: NDV-3 — 0.5mL injection IM
  Arms: NDV-3
Biological: Placebo — aluminum hydroxide and buffered saline
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study intended to assess the safety, tolerability and humoral and cellular immune response over a 12-month period after receiving one dose of either the NDV-3A vaccine, NDV-3 vaccine, or placebo. In addition, the clinical efficacy of NDV-3A vaccine in lowering the recurrence rate of vulvovaginal candidiasis (VVC) in patients with recurrent VVC (RVVC) will be evaluated relative to placebo.

DETAILED DESCRIPTION:
The purpose of the Phase 1b portion of this study is to compare the NDV-3A vaccine, the NDV-3 vaccine and the placebo head-to-head in the patient population of interest (women with RVVC) to evaluate safety and immunogenicity. The study size for comparing safety and immunogenicity (N=15 per group) is based on the dose comparison design used in study NDV3-001 (clinical trials.gov Identifier NCT01273922).

The primary purpose of the Phase 2a portion of this study is to further evaluate safety, tolerability, and immunogenicity of the NDV-3A vaccine compared to placebo in a patient population of interest (women with RVVC). The secondary purpose is to determine whether the NDV-3A vaccine decreases the recurrence rate of VVC in 18-50 year old women with RVVC when compared to placebo. The study size for evaluating efficacy (N=87 per group) is based on assuming a 50% rate of VVC recurrences over the 6 month post-vaccination period in the placebo group and a 50% vaccine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Has been informed of the nature of the study and has agreed to and is able to read, review, and sign the informed consent document prior to Screening.
* Is a female between 18-50 years of age, inclusive, at the time of vaccination on an acceptable form of birth control.
* Has a current episode of VVC (at Screening/Day -14) that can be confirmed with acute signs and symptoms of VVC (Composite Questionnaire score of ≥3) and a positive vaginal mycological culture for C. albicans.
* Has a history of 2 or more documented episodes of VVC in the 12 months prior to Screening, including at least one of the previous episodes confirmed by positive results from a diagnostic lab test specific for the presence of Candida. Additional episodes may be self-reported.
* Has a normal Papanicolaou (Pap) smear from the previous 12 months, or has no clinically significant abnormalities on a Pap smear taken at study entry as judged and documented by the investigator(s).
* Is in general good health as judged and documented by the investigator(s)

Exclusion Criteria:

* Reports receiving any systemic or topical vaginal antifungal therapy for 4 weeks prior to study entry.
* Mycological results from Study Day -14 or earlier cultures taken within 4 weeks prior to vaccination that show other yeast species (e.g., C. glabrata, C. tropicalis, etc.) as the cause of vaginitis.
* Has other active infectious cause(s) of vulvovaginitis (e.g., bacterial vaginosis, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhea, symptomatic Herpes Simplex Virus-1 (HSV-1), symptomatic HSV-2, or symptomatic human papilloma virus) at Screening or other vaginal or vulvar conditions that would confound the interpretation of clinical response as judged by the investigator(s).
* Will be under treatment or surgery at the start of the study for cervical intraepithelial neoplasia (CIN) or cervical carcinoma.
* Reports any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s), diagnosed diabetes mellitus (controlled or not) or psychiatric disease that would confound the interpretation of clinical response as judged by the investigator(s).
* Reports a history of allergic response(s) or other serious reactions to nickel, aluminum, or yeast products
* Reports a history of clinically significant allergies including food or drug allergies, anaphylaxis (or other serious reaction) to vaccines.
* Has a known history of or active infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Reports receiving or planning to receive any investigational drug, investigational vaccine, or investigational device within 4 weeks prior to vaccination, and at any other time during their participation in the study.
* Reports receiving or planning to receive any other live vaccine within 3 weeks prior to vaccination and for 3 weeks after vaccination.
* Reports having or shows evidence of a recent history of drug or alcohol abuse.
* Reports the use or planned use of any immunosuppressive drugs, including systemic or topical vaginal corticosteroids, within 4 weeks prior to vaccination, with the exception of topical steroids (e.g., Over-The-Counter hydrocortisone) used elsewhere on the body.
* Reports the use or planned use of any medications or treatments that may alter immune responses to the study vaccine within 3 weeks prior to vaccination
* Reports receiving any blood products within 3 months prior to vaccination and throughout the study.
* Reports donating blood/plasma within 4 weeks prior to vaccination.
* Is pregnant or intends to become pregnant over the course of the study, breastfeeding, or has any other medical and/or social (e.g., non-compliant) reason which, in the opinion of the investigator(s), would prevent participation in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hennessey, Jr., Ph.D., Study Director — NovaDigm Therapeutics, Inc.
Locations (20):
- United States (20):
  - Precision Trials LLC, Phoenix, Arizona
  - Arkansas Women's Center, Little Rock, Arkansas
  - Women's Health Care Research Corp, San Diego, California
  - McCann MD Research, Inc., Torrance, California
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - KO Clinical Research, LLC, Fort Lauderdale, Florida
  - Miami Clinical Research, LLC, Miami, Florida
  - Community Medical Research, Miami Beach, Florida
  - Community Medical Research LLC, North Miami, Florida
  - MedPharmics, Metairie, Louisiana
  - WSU Physician's Group, Detroit, Michigan
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Lawrence OB/Gyn Clinical Research, Lawrenceville, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Suffolk Ob/Gyn, Port Jefferson, New York
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Magnolia OB/GYN Research Center, LLC, Myrtle Beach, South Carolina
  - Advanced Research Associates, Corpus Christi, Texas
  - Discovery Clinical Trials- HCWC, LLC, Dallas, Texas
  - TMC Life Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Presentations at scientific meetings and publication

REFERENCES:
- [Derived] Edwards JE Jr, Schwartz MM, Schmidt CS, Sobel JD, Nyirjesy P, Schodel F, Marchus E, Lizakowski M, DeMontigny EA, Hoeg J, Holmberg T, Cooke MT, Hoover K, Edwards L, Jacobs M, Sussman S, Augenbraun M, Drusano M, Yeaman MR, Ibrahim AS, Filler SG, Hennessey JP Jr. A Fungal Immunotherapeutic Vaccine (NDV-3A) for Treatment of Recurrent Vulvovaginal Candidiasis-A Phase 2 Randomized, Double-Blind, Placebo-Controlled Trial. Clin Infect Dis. 2018 Jun 1;66(12):1928-1936. doi: 10.1093/cid/ciy185. PMID 29697768

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: aluminum hydroxide and buffered saline
  Placebo: 0.5 mL injection IM
Period: Overall Study
Arm/Group | Placebo | NDV-3A | NDV-3
Started | 85 | 89 | 14
Completed | 64 | 67 | 12
Not Completed | 21 | 22 | 2
Not completed — Lost to Follow-up | 7 | 6 | 0
Not completed — Physician Decision | 1 | 5 | 0
Not completed — Withdrawal by Subject | 9 | 9 | 2
Not completed — Non compliance or other reasons | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo: aluminum hydroxide adjuvant
  Placebo: 0.5 mL injection IM
- Total: Total of all reporting groups
Arm/Group | Placebo | NDV-3A | NDV-3 | Total
Number analyzed (Participants) | 85 | 89 | 14 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (8.80) | 32.1 (8.82) | 35.4 (10.70) | 32.5 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 89 | 14 | 188
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 36 | 3 | 66
  Not Hispanic or Latino | 58 | 53 | 11 | 122
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 17 | 19 | 2 | 38
  White | 64 | 68 | 12 | 144
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85 | 89 | 14 | 188

OUTCOME MEASURES:

1. Primary Outcome: Summary of Injection Site Reactions for the Safety Population Over the 12-months Post Vaccination Period
Description: Summary of injection site reactions for the safety population over the 12-months post-vaccination period in the NDV-3A vaccine group, the NDV-3 vaccine group, and the placebo group.
Time Frame: 12-month
Population: All enrolled patients.
Measure: Count of Units; unit: AEs
Units Other Than Participants: AEs
Arm/Group | Placebo | NDV-3A | NDV-3
Number analyzed (Participants) | 85 | 89 | 14
Number analyzed (AEs) | 279 | 358 | 31
AEs
  Patients with >= 1 injection site reaction | 72 | 79 | 10
  Induration | 25 | 46 | 0
  Pain | 56 | 70 | 7
  Redness | 34 | 45 | 2
  Swelling | 28 | 47 | 2
  Tenderness | 64 | 71 | 10

2. Secondary Outcome: Number of Patients <40 Years Old Who Were Recurrence-free Over the 12-month Post-vaccination Period
Description: Number of patients <40 years old with documented RVVC who were recurrence-free over the 12-month post-vaccination period in the NDV-3A vaccine group and the placebo group
Time Frame: 12 months
Population: Participants <40 years old
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo: aluminum hydroxide adjuvant
  Placebo: 0.5mL injection IM
Arm/Group | Placebo | NDV-3A
Number analyzed (Participants) | 50 | 57
Participants | 11 | 24
Statistical Analysis 1: Comparison: Placebo vs NDV-3A; Test type: Equivalence — The proportion of patients in each group was summarized with point estimates and their 95% confidence interval; p = 0.03, Wilcoxon (Mann-Whitney); Cox Proportional Hazard = 0.39, 95% CI 2-sided [0.17 to 0.91]

3. Secondary Outcome: Number of Patients Who Were Recurrence-free Over the 12-month Post-vaccination Period
Description: Number of patients with documented RVVC who were recurrence-free over the 12-month post-vaccination period in the NDV-3A vaccine group and the placebo group
Time Frame: 12 months
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NDV-3A
Number analyzed (Participants) | 68 | 74
Participants | 17 | 28
Statistical Analysis 1: Comparison: Placebo vs NDV-3A; Test type: Equivalence — The proportion of patients in each group was summarized with point estimates and their 95% confidence interval; p = 0.10, Wilcoxon (Mann-Whitney); Cox Proportional Hazard = 0.55, 95% CI 2-sided [0.27 to 1.13]

4. Secondary Outcome: Time to First VVC Episode From Study Day 17 to 360 - Participants <40 Years Old
Description: Time-to-onset of first VVC episode from Study Day 17 for the NDV-3A vaccine group and the placebo group
Time Frame: 12 months
Population: Participants < 40 years old
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | NDV-3A
Number analyzed (Participants) | 50 | 57
Days | 105 [45 to 325] | 210 [95 to 360]

5. Secondary Outcome: Time to First VVC Episode From Study Day 17 to 360 - All Participants
Description: Time-to-onset of first VVC episode from Study Day 17 for the NDV-3A vaccine group and the placebo group
Time Frame: 12 months
Population: All participants
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | NDV-3A
Number analyzed (Participants) | 68 | 74
Days | 135 [50 to 330] | 175 [70 to 350]

6. Secondary Outcome: Serum Anti-Als3 IgG Titers Over the 12-month Post-vaccination Period
Description: Serum anti-Als3 IgG titers will be measured by ELISA at pre-defined time points over the 12-month post-vaccination period in the NDV-3A vaccine group, the NDV-3 vaccine group, and the placebo group.
Time Frame: 0, 14, 28, 90, 180 and 360 days
Measure: Geometric Mean (Standard Deviation); unit: Titer (dilution^-1)
Arm/Group | Placebo | NDV-3A | NDV-3
Number analyzed (Participants) | 85 | 89 | 14
Titer (dilution^-1)
  Day 0 | 465 (3.3) | 434 (3.5) | 305 (3.1)
  Day 14 | 464 (3.6) | 37381 (3.9) | 18078 (4.6)
  Day 28 | 419 (3.3) | 31459 (3.6) | 13674 (4.6)
  Day 90 | 447 (3.2) | 17818 (3.5) | 10868 (3.8)
  Day 180 | 523 (3.5) | 10852 (3.5) | 6297 (3.9)
  Day 360 | 371 (3.6) | 5349 (3.2) | 4999 (3.9)

7. Secondary Outcome: Serum Anti-Als3 IgA1 Titers Over the 12-month Post-vaccination Period
Description: Serum anti-Als3 IgA1 titers will be measured by ELISA at pre-defined time points over the 12-month post-vaccination period in the NDV-3A vaccine group, the NDV-3 vaccine group, and the placebo group.
Time Frame: 0, 14, 28, 90, 180 and 360 days
Population: All participants
Measure: Geometric Mean (Standard Deviation); unit: Titer (dilution^-1)
Arm/Group | Placebo | NDV-3A | NDV-3
Number analyzed (Participants) | 85 | 89 | 14
Titer (dilution^-1)
  Day 0 | 937 (5.6) | 1011 (5.5) | 657 (3.1)
  Day 14 | 954 (6.4) | 63834 (5.1) | 44866 (3.7)
  Day 28 | 850 (5.5) | 43557 (5.2) | 30118 (3.2)
  Day 90 | 1062 (6.0) | 23053 (5.1) | 20349 (3.1)
  Day 180 | 982 (7.3) | 18215 (5.9) | 14633 (3.4)
  Day 360 | 563 (7.3) | 8727 (5.8) | 12357 (3.1)

8. Secondary Outcome: Cervicovaginal Wash Anti-Als3 IgG Titers Over the 12-month Post-vaccination Period
Description: Cervicovaginal wash anti-Als3 IgG titers will be measured by ELISA at pre-defined time points over the 12-month post-vaccination period in the NDV-3A vaccine group, the NDV-3 vaccine group, and the placebo group.
Time Frame: 0, 14, 28, 90, 180 and 360 days
Population: All participants
Measure: Geometric Mean (Standard Deviation); unit: Titer (dilution^-1)
Arm/Group | Placebo | NDV-3A | NDV-3
Number analyzed (Participants) | 85 | 89 | 14
Titer (dilution^-1)
  Day 0 | 2.03 (5.27) | 1.93 (4.19) | 1.47 (4.69)
  Day 14 | 1.93 (5.15) | 20.67 (6.28) | 8.01 (8.09)
  Day 28 | 1.44 (3.63) | 24.98 (6.97) | 9.88 (14.49)
  Day 90 | 1.40 (3.97) | 14.28 (6.16) | 5.28 (4.11)
  Day 180 | 1.66 (4.55) | 7.68 (6.73) | 2.72 (6.42)
  Day 360 | 1.44 (5.14) | 4.36 (6.39) | 2.76 (6.12)

9. Secondary Outcome: Cervicovaginal Wash Anti-Als3 IgA1 Titers Over the 12-month Post-vaccination Period
Description: Cervicovaginal wash anti-Als3 IgA1 titers will be measured by ELISA at pre-defined time points over the 12-month post-vaccination period in the NDV-3A vaccine group, the NDV-3 vaccine group, and the placebo group.
Time Frame: 0, 14, 28, 90, 180 and 360 days
Population: All participants
Measure: Geometric Mean (Standard Deviation); unit: Titer (dilution^-1)
Arm/Group | Placebo | NDV-3A | NDV-3
Number analyzed (Participants) | 85 | 89 | 14
Titer (dilution^-1)
  Day 0 | 4.86 (6.37) | 5.16 (5.38) | 2.02 (6.81)
  Day 14 | 4.99 (7.89) | 53.65 (7.00) | 28.24 (6.86)
  Day 28 | 3.44 (4.51) | 45.96 (8.56) | 22.22 (9.61)
  Day 90 | 2.87 (4.89) | 22.52 (7.50) | 5.75 (6.00)
  Day 180 | 3.13 (5.60) | 17.74 (5.76) | 10.17 (4.83)
  Day 360 | 3.39 (5.05) | 9.32 (7.06) | 5.02 (7.41)

10. Secondary Outcome: Als3-specific T-cell Production of Interferon Gamma Over the Post-vaccination Period
Description: Als3-specific T-cell production of interferon gamma will be measured by enzyme-linked immunospot (ELISpot) at pre-defined time points over the 12-month post-vaccination period in the NDV-3A vaccine group, the NDV-3 vaccine group, and the placebo group.
Time Frame: 0, 14, 90 days
Population: All participants
Measure: Geometric Mean (Standard Deviation); unit: Spot Forming Units
Arm/Group | Placebo | NDV-3A | NDV-3
Number analyzed (Participants) | 85 | 89 | 14
Spot Forming Units
  Day 0 | 2.7 (3.0) | 3.6 (3.3) | 2.6 (3.4)
  Day 14 | 3.0 (3.2) | 22.8 (5.3) | 22.1 (7.7)
  Day 90 | 3.2 (3.5) | 16.6 (4.6) | 15.1 (4.9)

11. Secondary Outcome: Als3-specific T-cell Production of Interleukin-17A Over the Post-vaccination Period
Description: Als3-specific T-cell production of interleukin-17A will be measured by enzyme-linked immunospot (ELISpot) at pre-defined time points over the 12-month post-vaccination period in the NDV-3A vaccine group, the NDV-3 vaccine group, and the placebo group.
Time Frame: 0, 14, 90 days
Population: All Participants
Measure: Geometric Mean (Standard Deviation); unit: Spot Forming Units
Arm/Group | Placebo | NDV-3A | NDV-3
Number analyzed (Participants) | 85 | 89 | 14
Spot Forming Units
  Day 0 | 3.4 (4.1) | 4.2 (4.4) | 5.2 (4.1)
  Day 14 | 2.6 (3.4) | 9.6 (5.3) | 11.1 (5.4)
  Day 90 | 2.9 (3.5) | 6.6 (3.9) | 3.3 (3.7)

ADVERSE EVENTS:
Time Frame: 12-months
Arm/Group | Placebo | NDV-3A | NDV-3
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/89 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/89 | 0/14
Other Adverse Events (participants affected / at risk) | 48/85 | 35/89 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | NDV-3A (N=89) | NDV-3 (N=14)
Anemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 15 | 13 | 1
Urinary tract infection (Infections and infestations) | 16 | 7 | 1
Nasopharyngitis (Infections and infestations) | 6 | 6 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 0
Headache (Nervous system disorders) | 4 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less